CLINICAL TRIAL: NCT03888469
Title: Clinical Comparison of DDT2 Contact Lens and a Daily Disposable Contact Lens - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-C007
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Refractive Error; Myopia
Keywords: Visual acuity; VA; Daily disposable contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DDT2, then 1DAVM (Other): Verofilcon A contact lenses worn first, with etafilcon A contact lenses worn second, as randomized. Each product was worn bilaterally (in both eyes) for 8 -1/+2 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Etafilcon A contact lenses
- 1DAVM, then DDT2 (Other): Etafilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each product was worn bilaterally (in both eyes) for 8 -1/+2 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Etafilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Investigational daily disposable soft contact lenses
  Other Names: DDT2
Device: Etafilcon A contact lenses — Commercially available daily disposable soft contact lenses
  Other Names: 1DAVM; 1-DAY ACUVUE® MOIST

SUMMARY:
The purpose of this study was to evaluate visual acuity at distance when wearing DDT2 contact lenses compared to Acuvue Moist contact lenses.

DETAILED DESCRIPTION:
Subjects were expected to attend 3 study visits and wear study lenses for approximately 14 - 20 days (7 - 10 days for each product).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Informed Consent Form that has been approved by an Institutional Review Board.
* Willing and able to attend all scheduled study visits as required per protocol.
* Current wearer of spherical soft contact lenses.

Key Exclusion Criteria:

* Any ocular condition that contraindicates contact lens wear.
* Previous or current habitual wearer of ACUVUE® MOIST or DAILIES TOTAL1® contact lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research
Locations (5):
- United States (5):
  - Alcon Investigative Site, Jacksonville, Florida
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Orlando, Florida
  - Alcon Investigative Site, Powell, Ohio
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 5 study centers in the United States (US).
Pre-assignment Details: This reporting group includes all randomized subjects (92).
Groups:
- DDT2, Then 1DAVM: Verofilcon A contact lenses worn first, with etafilcon A contact lenses worn second, as randomized. Each product worn bilaterally (in both eyes) for 8 -1/+2 days in a daily disposable modality.
- 1DAVM, Then DDT2: Etafilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each product worn bilaterally (in both eyes) for 8 -1/+2 days in a daily disposable modality.
Period: First Wear Period (8 -1/+2 Days)
Arm/Group | DDT2, Then 1DAVM | 1DAVM, Then DDT2
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0
Period: Second Wear Period (8 -1/+2 Days)
Arm/Group | DDT2, Then 1DAVM | 1DAVM, Then DDT2
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | DDT2, Then 1DAVM | 1DAVM, Then DDT2 | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (8.5) | 31.5 (7.8) | 32.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 44 | 38 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 40 | 83
  Black or African American | 2 | 4 | 6
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance Visual Acuity With Study Lenses
Description: Visual acuity was assessed and collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 8, each product
Population: Full Analysis Set (FAS): All randomized subjects who were exposed to any study lenses evaluated in this study, with the exception of the lenses used at Visit 1 for optimization and fitting.
Measure: Least Squares Mean (Standard Error); unit: logMar
Units Other Than Participants: eyes
Groups:
- DDT2: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
- 1DAVM: Etafilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
Arm/Group | DDT2 | 1DAVM
Number analyzed (Participants) | 92 | 92
Number analyzed (eyes) | 184 | 184
logMar | -0.13 (0.008) | -0.12 (0.008)
Statistical Analysis 1: Comparison: DDT2 vs 1DAVM; Test type: Non-Inferiority — Non-inferiority margin = 0.05; Mixed effects repeated measures model; Mixed effects repeated measures model with terms for lens, period and sequence as fixed effects and subject as a random effect; Least Squares Mean Difference = -0.00, 95% CI 1-sided [upper limit 0.00] — Difference = DDT2 - Moist

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent to study exit (approximately 14-20 days). The safety analysis set included all subjects/eyes exposed to any study lenses evaluated in this study, with the exception of the lenses used at Visit 1 for the purpose of parameter optimization and fitting, as they were not intended for the assessment of safety.
Description: Adverse events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population of ocular AEs is reported in units of eyes; all other populations are reported in units of subjects.
Groups:
- DDT2 - Ocular; DDT2 - Systemic / Nonocular: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
- 1DAVM - Ocular; 1DAVM - Systemic / Nonocular: Etafilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
Arm/Group | DDT2 - Ocular | DDT2 - Systemic / Nonocular | 1DAVM - Ocular | 1DAVM - Systemic / Nonocular
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/92 | 0/184 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/92 | 0/184 | 0/92
Other Adverse Events (participants affected / at risk) | 0/184 | 0/92 | 0/184 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03888469/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03888469/SAP_001.pdf